CLINICAL TRIAL: NCT04867278
Title: External Beam Radiotherapy as Prophylaxis for Heterotopic Ossification After Surgical Fixation of Acetabular Fractures: a Prospective, Randomized Feasibility Study
Brief Title: Heterotopic Ossification Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert O'Toole, Head of the UM SOM's Division of Orthopaedic Traumatology and Chief of Orthopaedic Traumatology and CHief of Orthopaedics for the University of Maryland Medical Center's (UMMS) R Adams Cowley Shock Trauma Center, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00093659
Record Dates: First submitted 2021-04-21; First posted 2021-04-30 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Acetabular Fracture; Heterotopic Ossification
MeSH Terms: conditions — Ossification, Heterotopic | interventions — Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Beam Radiation (XRT) with Debridement (Experimental): Patients will receive gluteus minimus debridement in the OR, which is the standard of care at Shock Trauma. If randomized to the treatment group, patients that undergo surgical fixation of an acetabular fracture via a posterior or combined anterior and posterior approach will undergo a single fraction of external beam radiotherapy to the surgical site within 72 hours of surgery. This treatment is currently the standard procedure performed for all patients who undergo a posterior or combined approach at our institution.
  Interventions: Procedure: External Beam Radiation (XRT); Procedure: Debridement
- Debridement Alone (Control) (Active Comparator): The control treatment arm will only include gluteus minimus debridement in the OR and will not receive XRT.
  Interventions: Procedure: Debridement

INTERVENTIONS:
Procedure: External Beam Radiation (XRT) — Patients that undergo surgical fixation of an acetabular fracture will receive debridement and a single fraction of external beam radiotherapy to the surgical site within 72 hours of surgery.
  Arms: External Beam Radiation (XRT) with Debridement
Procedure: Debridement — Gluteus minimus debridement in the OR

SUMMARY:
One complication that can occur after surgery on the acetabulum is the development of bone in abnormal places such as muscle and soft tissues. There is some evidence that a single dose of radiation to the surgical site within 3 days of surgery will prevent this abnormal bone from forming. However, there are no high quality studies proving that radiation works any better than doing nothing at all. The purpose of our study is to determine whether there is a difference in abnormal bone formation after acetabular surgery when patients are treated with external beam irradiation versus no treatment.

DETAILED DESCRIPTION:
Heterotopic ossification (HO) is a common complication after surgical fixation of acetabular fractures, with incidence rates reported as high as 90%. HO can be a debilitating complication and surgical excision for more severe cases carries a high complication rate. Numerous strategies have been employed to prevent HO formation but results are mixed and the optimal treatment strategy remains controversial.

The most common modalities used to prevent HO formation are oral administration of indomethacin or single-dose external beam irradiation therapy (XRT). Despite the common use of indomethacin and observational data to support its use, more recent randomized controlled trials (RCTs) have failed to demonstrate any significant reduction in the incidence of severe HO when patients were administered 6 weeks of indomethacin versus placebo. Similarly, XRT has been shown to be effective against HO formation in smaller observational studies, but there are no adequately powered RCTs to support its use compared to placebo.

Given the high incidence, impact on outcomes, and controversy regarding treatment, there remains a need for continued research to determine optimal treatment strategies for HO prophylaxis. While XRT remains standard of care for prophylaxis at many centers, including our own, there are no RCTs to support its use. Given the associated cost and resources, and potential risk even if minor, our study will help determine the feasibility of a larger RCT to help determine if the use of XRT is justified.

For this feasibility study, eligible patients will be randomized to XRT versus control. Both arms will receive gluteus minimus debridement in the OR, which is the standard of care at Shock Trauma. If randomized to the treatment group, patients that undergo surgical fixation of an acetabular fracture via a posterior or combined anterior and posterior approach will undergo a single fraction of external beam radiotherapy to the surgical site within 72 hours of surgery. This treatment is currently the standard procedure performed for all patients who undergo a posterior or combined approach at our institution. The control treatment arm will only include gluteus minimus debridement in the OR and will not receive XRT. We will have 30 patients randomized to each group. We will look at consent rate, power, and HO formation on 3 month post-op radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18+ with an acute acetabular fracture
* Indicated for surgical fixation via a posterior or combined anterior and posterior approach

Exclusion Criteria:

* Contraindication to radiotherapy such as history of cancer/RT
* Patients that are getting an acute total hip arthroplasty at the time of fixation of the acetabular fracture
* Not English speaking
* Not a Maryland resident or likely to have difficulty returning for post-op follow up(s) (i.e. homeless, incarceration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-05-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Shock Trauma Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sagi HC, Jordan CJ, Barei DP, Serrano-Riera R, Steverson B. Indomethacin prophylaxis for heterotopic ossification after acetabular fracture surgery increases the risk for nonunion of the posterior wall. J Orthop Trauma. 2014 Jul;28(7):377-83. doi: 10.1097/BOT.0000000000000049. PMID 24625922
- [Background] Matta JM, Siebenrock KA. Does indomethacin reduce heterotopic bone formation after operations for acetabular fractures? A prospective randomised study. J Bone Joint Surg Br. 1997 Nov;79(6):959-63. doi: 10.1302/0301-620x.79b6.6889. PMID 9393912
- [Background] Karunakar MA, Sen A, Bosse MJ, Sims SH, Goulet JA, Kellam JF. Indometacin as prophylaxis for heterotopic ossification after the operative treatment of fractures of the acetabulum. J Bone Joint Surg Br. 2006 Dec;88(12):1613-7. doi: 10.1302/0301-620X.88B12.18151. PMID 17159174
- [Background] Moore KD, Goss K, Anglen JO. Indomethacin versus radiation therapy for prophylaxis against heterotopic ossification in acetabular fractures: a randomised, prospective study. J Bone Joint Surg Br. 1998 Mar;80(2):259-63. doi: 10.1302/0301-620x.80b2.8157. PMID 9546456
- [Background] Burd TA, Lowry KJ, Anglen JO. Indomethacin compared with localized irradiation for the prevention of heterotopic ossification following surgical treatment of acetabular fractures. J Bone Joint Surg Am. 2001 Dec;83(12):1783-8. doi: 10.2106/00004623-200112000-00003. PMID 11741055

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | External Beam Radiation (XRT) With Debridement | Debridement Alone (Control)
Started | 59 | 58
Completed | 54 | 50
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | External Beam Radiation (XRT) With Debridement | Debridement Alone (Control) | Total
Number analyzed (Participants) | 54 | 50 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 49 | 101
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11) | 37 (13) | 36 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 35 | 40 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 53 | 48 | 101
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 29 | 65
  White | 16 | 19 | 35
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 50 | 104
Head Injury [Count of Participants; unit: Participants] | 11 | 10 | 21
Acetabular fracture dislocation [Count of Participants; unit: Participants] | 25 | 25 | 50
Associated fracture pattern [Count of Participants; unit: Participants] — Associated fracture patterns include the following: anterior with posterior hemitransverse, posterior-column with posterior-wall, and transverse with posterior-wall.
  Participants | 26 | 24 | 50
Surgical Approach: Kocher-Langenbeck [Count of Participants; unit: Participants] — The Kocher-Langenbeck approach is the method for the reduction and fixation of hip fractures that require fixation via a posterior approach.
  Participants | 49 | 44 | 93
Surgical Approach: Combined anterior and posterior [Count of Participants; unit: Participants] — A combined anterior and posterior surgical approach to the hip joint is a procedure that allows access to both the front and back of the hip joint. This approach is used for complex arthroplasty and reconstruction, and can be performed with minimal muscle release.
  Participants | 5 | 6 | 11
Trochanteric osteotomy [Count of Participants; unit: Participants] | 3 | 3 | 6
Gluteus minimus muscle debridement [Count of Participants; unit: Participants] | 51 | 49 | 100
NSAIDS for pain management [Count of Participants; unit: Participants] | 19 | 19 | 38
Closed suction drain at wound closure [Count of Participants; unit: Participants] | 22 | 20 | 42
Tranexamic acid used [Count of Participants; unit: Participants] | 14 | 20 | 34
Mechanical ventilation [Count of Participants; unit: Participants] | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe HO Formation
Description: Severe HO formation classified as Brooker class III-IV.
Time Frame: 3 months post-op
Measure: Count of Participants; unit: Participants
Arm/Group | External Beam Radiation (XRT) With Debridement | Debridement Alone (Control)
Number analyzed (Participants) | 54 | 50
Participants | 3 | 9

2. Secondary Outcome: Number of Participants With Any HO Formation
Description: Any HO formation classified as Brooker class I-IV.
Time Frame: 3 months post-op
Measure: Count of Participants; unit: Participants
Arm/Group | External Beam Radiation (XRT) With Debridement | Debridement Alone (Control)
Number analyzed (Participants) | 54 | 50
Participants | 10 | 17

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 3 months post-op for each patient.
Arm/Group | External Beam Radiation (XRT) With Debridement | Debridement Alone (Control)
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/50
Other Adverse Events (participants affected / at risk) | 2/54 | 3/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | External Beam Radiation (XRT) With Debridement (N=54) | Debridement Alone (Control) (N=50)
Superficial SSI (Infections and infestations) | 2 (2) | 2 (2) — Surgical Site Infection (SSI) categorized as superficial.
Deep SSI (Infections and infestations) | 0 (0) | 1 (1) — Surgical Site Infection (SSI) categorized as deep.

LIMITATIONS AND CAVEATS:
A limitation of the current study is the fourteen-patient crossover from the XRT treatment arm to no XRT. These 14 patients were randomized to the XRT group, but did not receive XRT at all, thus crossing over to the no XRT group. Additionally, although the sample size was adequately powered, there were a relatively few number of study events. Lastly, although the study is multicenter, it is only 2 centers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT04867278/Prot_SAP_000.pdf